CLINICAL TRIAL: NCT00198289
Title: A Phase IIa Dose Escalation Study to Assess Safety and Pharmacokinetics of Aurexis® in Cystic Fibrosis Subjects Chronically Colonized With Staphylococcus Aureus in Their Lungs
Brief Title: Aurexis® in Cystic Fibrosis Subjects Chronically Colonized With Staphylococcus Aureus in Their Lungs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: INH-AUR-004
Record Dates: First submitted 2005-09-09; First posted 2005-09-20 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Staphylococcus Aureus
Keywords: Cystic Fibrosis; Staphylococcus aureus; lungs
MeSH Terms: conditions — Staphylococcal Infections; Cystic Fibrosis

INTERVENTIONS:
Drug: Aurexis® (tefibazumab)

SUMMARY:
Patients who are at least 7 years old with stable Cystic Fibrosis who have Staphylococcus aureus in their Lungs will be enrolled into the study and receive one dose of Aurexis® intravenously on Study Day 1, and will be followed until Study Day 57. Aurexis is a humanized monoclonal antibody that is designed to combat Staphylococcus aureus.

The purpose of this study is to assess the safety and pharmacokinetic profile (concentration of Aurexis in blood and sputum) of Aurexis. Additionally, certain tests and measurements will be conducted to preliminarily determine if Aurexis demonstrates any benefit to these patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ages > 7 years old

  * Diagnosis of CF as evidenced by sweat chloride test and/or genetic mutation testing
  * Sputum SA CFUs > 10,000 per mL
  * Ability to expectorate sputum
  * Ability to tolerate nasal lavage and collection of breath condensate
  * Willing to practice reliable birth control measures during the entire study period, if subject is of childbearing potential
  * Informed consent obtained from subject or legal guardian, and assent if appropriate

Exclusion Criteria:

* Burkholderia cepacia in sputum

  * Subjects who have had changes to their treatment regimen for CF in the past 6 weeks

    * Subjects can be screened 6 weeks after IV antibiotic completion
    * Subjects can be screened 7 days after oral antibiotic completion
  * Received an investigational drug within 30 days of study entry
  * Received any immune globulin or blood product within 30 days of study entry
  * History of hypersensitivity to immune globulin preparations
  * Undergoing any type of dialysis or expected to start dialysis within 30 days
  * Pregnant or nursing females
  * Considered unlikely to comply with the study procedures or to return for scheduled post-treatment evaluations

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2005-04; Study Completion 2006-06

PRIMARY OUTCOMES:
To evaluate the safety of a single dose of Aurexis® in stable subjects with CF who are chronically colonized with SA in their lungs
To evaluate the pharmacokinetics of a single dose of Aurexis® in stable subjects with CF who are chronically colonized with SA in their lungs

SECONDARY OUTCOMES:
To evaluate the biologic and clinical effects of a single dose of Aurexis® in stable subjects with CF who are chronically colonized with SA in their lungs on:
Changes in bacterial load of SA in sputum as determined by colony counts
Changes in inflammatory mediators in nasal lavage fluid, breath condensate and plasma, including IL-1β, IL-6, IL-8, and TNFα.
Changes in oxidant/antioxidant balance in nasal lavage, breath condensate and plasma including GSH, GSSG, redox potential, cysteine, and cystine
Changes in pulmonary function tests as determined by FVC, FEV1, and FEF25-75%

CONTACTS AND LOCATIONS:
Overall Officials: Seth Hetherington, M.D., Study Director — Inhibitex
Locations (1):
- Emory University, Atlanta, Georgia, United States